CLINICAL TRIAL: NCT01099787
Title: Pediatric Alliance for International Neurogastrointestinal Functional Research Registry
Brief Title: Pediatric Alliance for International Neurogastrointestinal Functional Research
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Carlo Di Lorenzo, Professor of Clinical Pediatrics, Nationwide Children's Hospital
Other Study IDs: IRB10-00022
Record Dates: First submitted 2010-04-07; First posted 2010-04-08 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- FAP IBS

SUMMARY:
To explore the predictive value of alarm signs ("red flags") for a diagnosis of functional gastrointestinal disorders (FGID) in children.

To assess the natural history of pain predominant functional gastrointestinal disorders (FGID) in newly diagnosed pediatric patients.

To document the benefit of various treatment regimens currently employed in managing FGID.

To assess the short- and long-term impact of various FGID regimens.

To allow physicians to gain a better understanding of the epidemiology of FGID.

Hypothesis:

There are presenting symptoms or results from diagnostic tests that are more likely to associated with conditions different from FAP or IBS.

Symptoms of children with FAP/IBS change overtime regardless of the treatments used.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 4 through 16 years of age (up to the day of the 17th birthday)
* Presenting with chronic or intermittent abdominal pain of any severity lasting at least 2 months may participate in the Registry.

Exclusion Criteria:

* Subjects age 10 and above will be asked to complete the questionnaire themselves. Those unable to complete the questionnaire (with only some help) should not be enrolled.
* Patients unable to participate in the program for at least 3 years should not be enrolled (i.e., anticipated move, etc.)

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients ages 4 through 16 years of age (up to the day of the 17th birthday) will be recruited from the Nationwide Children's Hospital Gastrointestinal Department that are presenting with chronic or intermittent abdominal pain of any severity lasting at least 2 months.
Sampling Method: Non-Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Di Lorenzo, M.D., Principal Investigator — Nationwide Children's Hospital
Locations (7):
- United States (6):
  - Connecticut Children's Hospital, Hartford, Connecticut
  - Childrens Memorial Hospital, Chicago, Illinois
  - LSU Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital Boston, Boston, Massachusetts
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Emma Children's Hospital, Amsterdam, Netherlands